CLINICAL TRIAL: NCT05928208
Title: The Role of Point-of-care Polymerase Chain Reaction in Managing Nosocomial Pneumonia
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Balan Andrei Mihai, MD, Phd student, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: 82/03.03.2017
Record Dates: First submitted 2017-06-18; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Nosocomial Pneumonia
Keywords: polymerase chain reaction
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: no intervention — no intervention

SUMMARY:
The study compares a device that is used for the detection of bacteria and MDR pathogens from skin, soft tissue and nose with the gold-standard (microbiological lab). It is a novel use for this device because it has been used in samples from the lower-respiratory tract.

DETAILED DESCRIPTION:
The purpose of this study is to find out if a POC-PCR device can be use in the diagnosis of hospital acquired pneumonia and ventilation-associated pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* patients that are admitted for at least 48 hours
* radiological findings typical for pneumonia
* signs of infection

Exclusion Criteria:

* patient or patient relatives doesn't accept to enter the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with symptoms of nosocomial pneumonia
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
To determine the sensibility and specificity of the device GeneXpert in diagnosis of pneumonia | 4 years
  Comparison between device and gold standard
Utility of POC-PCR in managing pneumonia | 4 years
  Decision making in pneumonia management

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Balan, MD, Principal Investigator — Universitatea de Medicina si Farmacie "Iuliu Hatieganu" Cluj-Napoca
Locations (1):
- Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No